CLINICAL TRIAL: NCT03506607
Title: Exercise Training Under Hypoxic Conditions in Lower Extremity Artery Disease
Brief Title: Hypoxic Exercise in Lower Extremity Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Lucia Mazzolai, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017_00397_Phase1
Record Dates: First submitted 2018-03-28; First posted 2018-04-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Peripheral Arterial Disease
Keywords: exercise; cardiovascular; normobaric hypoxia
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise in hypoxia 1500m (Experimental): During this visit, subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). The ambient air will be mixed with nitrogen and inspired oxygen fraction will be reduced to 16%.
  Interventions: Other: Exercise in hypoxia 1500m
- Exercise in hypoxia 2500m (Experimental): During this visit, subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). The ambient air will be mixed with nitrogen and inspired oxygen fraction will be reduced to 14%.
  Interventions: Other: Exercise in hypoxia 2500m
- Exercise in normoxia (Placebo Comparator): During this visit, subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). For the exercise performed in normoxia conditions, subjects will breathe room air.
  Interventions: Other: Exercise in normoxia

INTERVENTIONS:
Other: Exercise in hypoxia 1500m — Subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). The ambient air will be mixed with nitrogen and inspired oxygen fraction will be reduced to 16%. The first 3 min will be performed at 70% of the mean speed calculated during a previous visit, and the last 3 min at an intensity between 12-14 on the Borg's scale.
  Arms: Exercise in hypoxia 1500m
Other: Exercise in hypoxia 2500m — Subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). The ambient air will be mixed with nitrogen and inspired oxygen fraction will be reduced to 14%. The first 3 min will be performed at 70% of the mean speed calculated during a previous visit, and the last 3 min at an intensity between 12-14 on the Borg's scale.
  Arms: Exercise in hypoxia 2500m
Other: Exercise in normoxia — Subjects will perform a 6-min treadmill exercise wearing an oronasal mask connected (through a hose) with a three-way valve to an altitude simulation device (Altitrainer; SMTech, Nyon, Switzerland). For the exercise performed in normoxia conditions, subjects will breathe room air. The first 3 min will be performed at 70% of the mean speed calculated during a previous visit, and the last 3 min at an intensity between 12-14 on the Borg's scale.
  Arms: Exercise in normoxia

SUMMARY:
The aim of this randomized controlled trial is to:

Phase I: To explore, in a first pilot phase, the adequate combination of hypoxia severity and exercise intensity in patients with symptomatic lower extremity artery disease (LEAD). Acute walking performances and physiological responses (vascular and muscular) to a normobaric hypoxic exercise performed will be assessed at two different altitudes (1500 m and 2500 m).

DETAILED DESCRIPTION:
The results of this first phase will then be used to determine the optimal hypoxic level for the exercise training program which will be assessed during the Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic LEAD (Fontaine stage ≥ IIa)
* ABI ≤ 0.9
* TBI ≤ 0.6 if incompressible arteries (diabetes and renal insufficiency)
* Signed written informed consent form

Exclusion Criteria:

* Neurological and neuromuscular disorders which can limit balance and walking
* Any history of altitude-related sickness
* Any health risks (assessed during clinical history) linked to hypoxia exposure
* Acclimatization or exposure to hypoxia of more than 2000 m for more than 48 h during a period of 6 months before the study
* Medication required for the treatment of migraines, claustrophobia that may interfere with the interpretation of the results
* Obstructive sleep apnea (> 25 Apnea-Hypopnea Index)
* Prior leg/foot amputation
* Pregnant women
* Cardiac contraindication to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Walking performance | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Total walking distance (in meters) during the 6 min treadmill test
Pain free walking time | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Pain free walking time during the 6 min treadmill test
Muscle oxygenation during exercise | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Muscle oxygenation during the 6 min treadmill test (assessed by near-infrared spectroscopy)
Pulse wave velocity | Before and after each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Pulse wave velocity before and after the 6 min treadmill test
Flow-mediated dilation | Before and after each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Flow-mediated dilation before and after the 6 min treadmill test
Pulse oxygen saturation | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Pulse oxygen saturation during the 6 min treadmill test

SECONDARY OUTCOMES:
Ankle-brachial index | Before and after each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Ankle-brachial index before and after the 6 min treadmill test
Toe-brachial index | Before and after each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Toe-brachial index before and after the 6 min treadmill test
Rate of perceived exertion | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Rate of perceived exertion (RPE) will be assessed using Borg's scale. RPE is a widely used and reliable indicator to monitor and guide exercise intensity. The scale allows individuals to subjectively rate their level of exertion during 6 min treadmill test. Patients will classify their RPE between 6 (light) and 20 (maximal).
Leg pain | After each 6 min treadmill test performed under hypoxic condition (1500 and 2500 m) and under normoxic condition (i.e., average of 3 weeks; one condition per week)
  Leg pain during exercise will be measured with a 10-points (0: "no pain" and 10: "worst imaginable pain") visual analogic scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Mazzolai, Prof, Principal Investigator — Division of angiology, Lausanne University Hospital
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No